

## Assent to Participate in Research (7 to 11 years of age)

## **BMT CTN 2207**

A Phase II Trial of Non-Myeloablative Conditioning and Transplantation of Haploidentical Related, Partially HLA-Mismatched, or Matched Unrelated Bone Marrow for Newly Diagnosed Patients with Severe Aplastic Anemia

| Subject's Name: | Date: |
|-----------------|-------|

- 1. Dr (s). [insert Dr (s) names here] is/are doing a research study about aplastic anemia.
- 2. We are asking you to take part in this research because we want to learn more about transplants and how well it works for your aplastic anemia.
- 3. If you agree to be in this study, you will be asked to:
  - Receive the transplant
  - Receive medicine to help with the transplant
  - Have tests to see how your body is doing. You will have these tests every few weeks or months for up to 1 year.
  - We will also ask you how you are feeling and how well you are able to do the things you normally do each day.

## When you are in a research study, sometimes good things and bad things can happen:

- 4. Things that happen to people in research studies that make them feel bad are called "risks." The risk (s) for this research study are:
  - Your body reacting to the transplant or the medicines to help with your transplant which may or may not occur. They could vary from mild, to medium, to serious, and you will be given medicine to help take care of it.
  - You could feel uncomfortable, afraid, lonely, or hurt. You can stop the study at any time you want to.

- Sometimes, the questions we ask can make you feel embarrassed or uncomfortable. You do not need to answer any questions you do not want to.
- You may get a bruise and feel some pain when we are drawing blood. Some of the blood can be saved for testing in the future. It will be drawn when other blood is being taken. You do not have to allow this extra blood to be drawn to be on the study.

These things may or may not happen to you. Some things may happen that the doctors do not know about yet.

- 5. Things that happen to people in research studies that are good are called "benefits." The benefit(s) for this research study are:
  - This study might help you need less treatment for your aplastic anemia.
- 6. We will do everything possible to keep your information private.
- 7. You do not have to be in this study if you do not want to. You may stop being in this study at any time- Remember, being in this study is up to you.
- 8. Please talk with your parent (s) or caregiver before you decide to be in this study. We will also ask your parent (s) or caregiver to give their permission for you to take part in this study. But even if they say "yes," you can still decide not to do this. Your doctor will still take care of you if you decide not to be in this study.
- 9. You can ask any questions that you have about the study. If you have other questions later, you can call your care team and doctor when next you see them.



[insert number (s) here

Sign your name on the line below if you agree to be in this study. You can also let us know if you want to allow us to take extra blood from you. Remember, you can change your mind at any time. You can keep a copy of this form at home.

## Minor Assent

| Print Name of Minor | <br>Age of Minor |
|-------------------------------------------|----------------------|
| Minor's Signature | Date |
| □ No, you may not take extra blood fr | om me for the future |
| □ No very many materials arrive blood for | and the faction |
| ☐ Yes, you may take extra blood from | me for the future. |